CLINICAL TRIAL: NCT03072030
Title: 01 - GamEvac-Combi-2016 " International Multicenter Study of the Immunogenicity of Medicinal Product GamEvac-Combi - Combined Vector-Based Vaccine Against Ebola Virus Disease, 0.5 ml+0.5 ml/Dose "
Brief Title: International Multicenter Study of the Immunogenicity of Medicinal Product GamEvac-Combi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: CREMS (Centre de Recherche Epidémiologie, Microbiologie et Soins médicaux ) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01 - GamEvac-Combi-2016; http://grls.rosminzdrav.ru (Registry Identifier: the Ministry of Health of the Russian Federation)
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-07

CONDITIONS: Ebola Virus Disease; Prevention
Keywords: Ebola Virus Disease; Hemorrhagic Fever, Ebola; Vaccines; GP protein, Ebola virus; Ebola Virus Vaccines
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: This clinical trial is designed as a double blind randomized placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Drug Group (Experimental): 1900 volunteers will be immunized with vaccine GamEvac-Combi They will receive product twice according to the following dosing regimen: on Day 1 (component A) and Day 21 of the study (component B) in the dose of 0.5 ml
  Interventions: Biological: GamEvac-Combi (vaccine)
- Placebo Drug Group (Placebo Comparator): 100 volunteers will be immunized with placebo They will receive product twice according to the following dosing regimen: on Day 1 (placebo - component A) and Day 21 of the study (placebo- component B) in the dose of 0.5 ml
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GamEvac-Combi (vaccine) — vaccination
  Arms: Active Drug Group
Biological: Placebo — vaccination
  Arms: Placebo Drug Group

SUMMARY:
The purpose of this study is to evaluate immunogenicity, epidemiological efficacy and safety of medicinal product GamEvac-Combi - Combined Vector-Based Vaccine against Ebola Virus Disease, 0.5 ml+0.5 ml/dose

DETAILED DESCRIPTION:
This clinical trial is designed as a double blind randomized placebo-controlled study to evaluate immunogenicity of medicinal product GamEvac-Combi - Combined Vector-Based Vaccine against Ebola Virus Disease, 0.5 ml+0.5 ml/dose.

The study includes three periods: screening, administration of the investigated product and follow-up. Vaccine will be administered to groups of volunteers (each group will include not more than 40 volunteers at a time; a new group of volunteers cannot be hospitalized before the earlier vaccinated volunteers are discharged from the hospital. In total, 8 visits will be held, including a screening visit; two of the visits will take place during the inpatient stage and six - during the outpatient observation.

Study design in the both facilities will be the same for all volunteers, except that the biomaterial collected for immunogenicity evaluation from volunteers included in the study in the Russian Federation will be delivered directly to the testing laboratory; biomaterial from volunteers included in the study in the Republic of Guinea will undergo primary specimen processing, be frozen and stored under the assigned temperature conditions in the research center and, as biomaterial is accumulated, it will be transported in a fridge to the study site.

In addition, laboratory tests for such concomitant infectious diseases, as yellow fever, Denge fever, Ebola and Marburg virus diseases will be carried out for epidemiological indications (i.e. in the endemic regions if disease cases are reported).

ELIGIBILITY:
Inclusion Criteria:

* Males and females within the age range from 18 to 60 years;
* written informed consent;
* absence of acute infectious diseases/relapses of chronic diseases at the time of vaccine administration and 7 days prior to the vaccination;
* absence of severe allergic diseases in the medical history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum disease)
* no serious post-vaccination complications in patient's history following the earlier administration of immunobiological products
* negative blood or urine test for pregnancy (for child-bearing age females) not more than 24 hours prior to the administration of the first dose of investigated product;
* absence of concomitant illnesses, especially dangerous or endemic for a particular region, proved by laboratory and/or clinical methods (malaria, yellow fever, Denge fever, Ebola or Marburg virus disease, poliomyelitis).
* negative results of HIV, hepatitis B and C and syphilis tests.
* adequate contraception for females and males of reproductive age.
* negative results of urine test for narcotic drug residues;
* negative result of breath alcohol test (in the expired air sample)
* absence of haematological malignancies
* absence of malignant neoplasms

Exclusion Criteria:

* - volunteer involvement in another study over the last 90 days;
* any immunization with vaccine over the last 30 days;
* symptoms of acute respiratory diseases within the last 7 days;
* administration of immunoglobulins or other blood products; taking immunosuppressive medications and/or immunomodulating agents over the last 3 months;
* pregnancy or breast feeding;
* exacerbation of allergic diseases, previous history of anaphylactic reactions or angioneurotic edema;
* previous history of hypersensitivity or allergic reactions to the administration of any vaccines;
* allergic reactions to the vaccine components;
* presence of a concomitant illness which might affect the evaluation of study results: active tuberculosis form, chronic liver and kidney diseases, serious thyroid dysfunction or other endocrine disorders (diabetes mellitus), severe hematopoietic diseases, epilepsy and other CNS disorders, myocardial infarction in the medical history, myocarditis, endocarditis, pericarditis, ischemic heat disease and other illnesses which, in opinion of the investigator, make patient ineligible for study enrollment or may affect the course of the study.
* blood donation (450 ml or more of blood or plasma) less than 2 months prior the study commencement date.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
determination of immunity duration by ELISA method | the total Time Frame is 12 month after the vaccination
  immunity duration determination by ELISA method includes time points in which the assessment of the immunity response (antibody titer) should be provided (21, 28, 42 days and 3, 6, 12 months after the vaccination respectively)

SECONDARY OUTCOMES:
assessment of antigen-specific cell-mediated immune response | on days 0 and 28
  determination of specific T-cell- mediated response to Ebola virus proteins vs. baseline values and placebo
determination of immunity duration in virus neutralization reaction | on days 0 and 42
  Determination of the immunity duration will be provided by the assessment of the neutralizing antibody titer for a virus in virus neutralization reaction vs. baseline values and placebo

OTHER OUTCOMES:
safety and tolerability | through study completion, an average of 1 year
  Incidence in the healthy volunteers vital parameters changes and the occurrence of systemic and local post-vaccination reactions in comparison with placebo; reviewing its impact on the vital parameters in healthy volunteers (systolic and diastolic blood pressure, heart rate, respiration rate, body temperature) and the occurrence of systemic and local post-vaccination reactions in comparison with placebo
epidemiological effectiveness of vaccination | through study completion, an average of 1 year"
  2. Where possible, to evaluate epidemiological effectiveness of vaccination based on the follow-on morbidity indicators of immunized and non-immunized individuals, manifestations of the epidemiological process in time and space

CONTACTS AND LOCATIONS:
Overall Officials: Sylla Ali Lathyr, Principal Investigator — physician administrator; Marina Rusanova, MD, PhD, Principal Investigator — doctor of infectious department
Locations (2):
- Centre de recherche en épidémiologie, microbiologie et de soins médicaux (CREMS) de Pastoria à Kindia, Kindia, Guinea
- Infectious Disease Clinical Hospital No. 1 of the Moscow Healthcare Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Logunov DY, Dolzhikova IV, Boiro MY, Kovyrshina AV, Dzharullaeva AS, Erokhova AS, Grousova DM, Tukhvatulin AI, Izhaeva FM, Simakova YV, Ordzhonikidze MK, Lubenets NL, Zubkova OV, Scheblyakov DV, Esmagambetov IB, Shmarov MM, Semikhin AS, Tukhvatulina NM, Shcherbinin DN, Tutykhina IL, Prokhorov GS, Khovaev AA, Demidova TN, Malishev NA, Merkulova LN, Voronina OL, Fedyakina IT, Kisteneva LB, Kolobukhina LV, Mishin DV, Elakov AL, Ermolova EI, Krasnoslobodtsev KG, Larichev VF, Kruzhkova IS, Burmistrov EM, Sheremet AB, Tokarskaya EA, Gromov AV, Reshetnikov DA, Fisun AI, Kotiv BN, Ovchinnikov DV, Ivchenko EV, Zhdanov KV, Zakharenko SM, Solovev AN, Ivanov AM, Sukachev VS, Gudkov RV, Maltsev OV, Gabdrakhmanov IA, Barsukov AV, Vashchenkov VV, Demianenko NI, Ignatev SB, Asiamov KV, Kirichenko NN, Liubimov AV, Volkov II, Kriukov EV, Bazarnov NK, Kolodiazhnaia VA, Kolomoets EV, Syromyatnikova SI, Chifanov DE, Andrus AF, Kutaev DA, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of GamEvac-Combi, a heterologous rVSV- and rAd5-vectored Ebola vaccine: a randomized controlled multicenter clinical trial in the Republic of Guinea and Russia. Front Immunol. 2025 Mar 20;16:1487039. doi: 10.3389/fimmu.2025.1487039. eCollection 2025. PMID 40207235